CLINICAL TRIAL: NCT04138979
Title: Intestinal Microbiota of Breast Cancer Patients Undergoing Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yunwei Wei 2019-09-13
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-09

CONDITIONS: Microbiota
Keywords: gut microbiota; 16S rRNA gene; breast cancer chemotherapy
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: 20 healthy volunteers were included in the healthy control group
- Disease group: First chemotherapy for breast cancer
  Interventions: Drug: cyclophosphamide

INTERVENTIONS:
Drug: cyclophosphamide — First use of chemotherapy after breast cancer
  Groups: Disease group

SUMMARY:
To date, few studies have addressed the link between gut microbiota and breast cancer chemotherapy, and previous studies have only provided a link between the gut and breast cancer.

DETAILED DESCRIPTION:
To date, few studies have addressed the link between gut microbiota and breast cancer chemotherapy, and previous studies have only provided a link between the gut and breast cancer.At present, studies on the interaction mechanism between intestinal flora and breast cancer mainly focus on two aspects: first, intestinal flora affects the occurrence and progress of breast cancer by affecting estrogen metabolism;Second, intestinal flora can influence the occurrence and treatment of breast cancer by affecting the regulation of the immune system.However, the specific types (or groups) of bacteria that promote the occurrence, development and mechanism of breast cancer still need to be further studied.In addition, since most of the current clinical studies on microorganisms and breast cancer are small sample studies, the accuracy of their conclusions remains to be studied.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* First use of chemotherapy after breast cancer

Exclusion Criteria:

* Pregnancy
* Lactation
* Cigarette smoking
* Alcohol addiction
* Hypertension
* Diabetes mellitus
* Lipid dysregulation
* BMI > 27
* Recent (< 3 months prior) use of antibiotics, probiotics, prebiotics, symbiotics, hormonal medication, laxatives, proton pump inhibitors, insulin sensitizers or Chinese herbal medicine
* History of disease with an autoimmune component, such as MS, rheumatoid arthritis, IBS, or IBD
* History of malignancy or any gastrointestinal tract surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients were included according to the inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Transcriptional changes in gut microbiota | baseline,1 day,7 day,14 days,22 days,29 days,36 days,44days,51days,58days,66days,73days,80days
  The microbiota measured by 16S rRNA gene

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luu TH, Michel C, Bard JM, Dravet F, Nazih H, Bobin-Dubigeon C. Intestinal Proportion of Blautia sp. is Associated with Clinical Stage and Histoprognostic Grade in Patients with Early-Stage Breast Cancer. Nutr Cancer. 2017 Feb-Mar;69(2):267-275. doi: 10.1080/01635581.2017.1263750. Epub 2017 Jan 17. PMID 28094541
- [Background] Qin J, Li R, Raes J, Arumugam M, Burgdorf KS, Manichanh C, Nielsen T, Pons N, Levenez F, Yamada T, Mende DR, Li J, Xu J, Li S, Li D, Cao J, Wang B, Liang H, Zheng H, Xie Y, Tap J, Lepage P, Bertalan M, Batto JM, Hansen T, Le Paslier D, Linneberg A, Nielsen HB, Pelletier E, Renault P, Sicheritz-Ponten T, Turner K, Zhu H, Yu C, Li S, Jian M, Zhou Y, Li Y, Zhang X, Li S, Qin N, Yang H, Wang J, Brunak S, Dore J, Guarner F, Kristiansen K, Pedersen O, Parkhill J, Weissenbach J; MetaHIT Consortium; Bork P, Ehrlich SD, Wang J. A human gut microbial gene catalogue established by metagenomic sequencing. Nature. 2010 Mar 4;464(7285):59-65. doi: 10.1038/nature08821. PMID 20203603